CLINICAL TRIAL: NCT05883592
Title: A Real-World Study on Distal Aortic Remodeling for Stanford Type B Aortic Dissection With Fabulous Thoracic Aortic Stent System
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hangzhou Endonom Medtech Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: Fabulous WQ-F01
Record Dates: First submitted 2023-05-18; First posted 2023-06-01 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Aortic Dissection
Keywords: Stent Graft
MeSH Terms: conditions — Aortic Dissection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fabulous Thoracic Aortic Stent System
  Interventions: Device: Fabulous Thoracic Aortic Stent System

INTERVENTIONS:
Device: Fabulous Thoracic Aortic Stent System — Endovascular treament in patients with aortic dissection with Fabulous Thoracic Aortic Stent System

SUMMARY:
To evaluate aortic remodeling of Fabulous thoracic aortic stent system in the treatment of acute and subacute Stanford type B aortic dissection (the changes of aortic diameter, cross-sectional area,and volume of true lumen, false lumen and total aorta in different aoritc levels, and false lumen thrombosis in different aoritc levels), and splanchnic artery perfusion.

DETAILED DESCRIPTION:
Fabulous Thoracic Aortic Stent System is specially designed for aortic dissection based on PETTICOAT technique.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old, regardless of gender;
2. Fabulous thoracic aortic stent System is suitable for the treatment of acute or subacute Stanford type B dissection, and the lesions meet one of the following criteria:

   1. It is necessary to treat distal lesions due to the presence of distal tears;
   2. The dissection involved a wide range, and there was collapse of the distal true cavity;
   3. Dissection combined with poor perfusion of distal branch vessels.
3. With appropriate arterial access and suitable for endovascular aortic repair;
4. Subjects could understand the purpose of the trial, volunteered to participate in the study, signed the informed consent form by themselves or their legal representatives, and were willing to complete the follow-up as required by the protocol.

Exclusion Criteria:

1. Patients have participated in clinical trials of other drugs or medical devices related to target lesion treatment or have participated in clinical trials of other drugs or medical devices and have not reached the primary endpoint;
2. Patients were unable or unwilling to participate in the study;
3. Patients were judged by the investigator to be ineligible for participation in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Stanford type B aortic dissection are treated with Fabulous Thoracic Aortic Stent System in the real world.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Change of diameter | 3 months, 6 months,12 months after operation
  The changes of true lumen, false lumen and total aortic diameter before and after surgery in the level of pulmonary artery bifurcation/left atrial (L1), the distal end of covered stent (L2), superior mesenteric artery (L3) and abdominal aortic bifurcation (L4) were recorded.
Changes of cross-sectional area | 3 months, 6 months,12 months after operation
  The changes of true lumen, false lumen and total aortic cross-sectional area before and after surgery in the level of pulmonary artery bifurcation/left atrial (L1), the distal end of covered stent (L2), superior mesenteric artery (L3) and abdominal aortic bifurcation (L4) were recorded.
Volumetric change | 3 months, 6 months,12 months after operation
  The volumes of the true lumen and false lumen of the aorta before and after surgery were measured from the covered stent placement segment, the proximal end of the bare stent to the level of celiac trunk, from the level of celiac trunk to the level of low kidney, and from the level of low kidney to the abdominal aorta bifurcation.

SECONDARY OUTCOMES:
Splanchnic arteries perfusion | 3 months, 6 months,12 months after operation
  The change rate of postoperative true lumen diameter of branch artery = (postoperative true lumen diameter - preoperative true lumen diameter)/preoperative true lumen diameter ×100%
Incidence of distal new entry | 3 months, 6 months,12 months after operation
  The number of visceral artery segment tears and infrarenal abdominal aorta segment tears were evaluated.
Tortuosity of the descending thoracic aorta | 3 months, 6 months,12 months after operation
  Tortuosity of the descending thoracic aorta = the length of left subclavian artery to descending aorta of coeliac trunk along the center lumen line/the outer curvature length of left subclavian artery to coeliac trunk
Immediate technical success | Immediate during surgery
  Immediate technical success was defined as the stent was successfully delivered to the intended site and released.
Incidence of type I and III endoleak | Immediate during surgery,3 months, 6 months,12 months after operation
Major adverse events occurring within 30 days after surgery | within 30 days after operation
  Refers to all-cause mortality, myocardial infarction, ischemic stroke or respiratory failure occurring within 30 days after surgery. More specifically, myocardial infarction refers to a drastic reduction or complete interruption of the coronary blood supply due to coronary artery disease, resulting in severe and prolonged acute ischemia of the corresponding myocardium, leading to necrosis of cardiomyocytes. Ischemic stroke refers to the end result of necrosis of brain tissue caused by narrowing or occlusion of the arteries supplying blood to the brain or insufficient blood supply to the brain. Respiratory failure is defined as a state resulting in significantly prolonged intubation, tracheotomy, deterioration of lung function, or other fatal outcomes.
Incidence of severe adverse events | 3 months, 6 months,12 months after operation
  Refers to an event that occurs during the clinical trial that results in mortality or serious deterioration in patient health, including a fatal illness or injury, a permanent defect in body structure or body function, or an event that requires medical or surgical intervention to avoid one or more permanent defects in body structure or body function.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing

IPD SHARING:
Plan to Share IPD: No